CLINICAL TRIAL: NCT06083207
Title: A Phase I/II, Multicenter, Open-label, First-in-human Study of IBI3003 in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of IBI3003 in Subjects With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIBI3003A101
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI3003 (Experimental)
  Interventions: Drug: IBI3003

INTERVENTIONS:
Drug: IBI3003 — Subjects will receive IBI3003 on Day 1 in a 28-day cycle (or intervals determined by the Investigator and Sponsor based on safety, toxicity and pharmacokinetic(PK) data), until death, disease progression, intolerable toxicity, start of a new anticancer treatment, withdrawal of consent for study participation, end of the study, or for a maximum of 24 months, whichever occurs first.

SUMMARY:
This is a phase 1/2 multicenter, open-label, first-in-human study of IBI3003. It includes a phase 1 dose escalation and expansion section to identify maximum tolerated dose(MTD)/recommended Phase 2 Dose(RP2D) of IBI3003, plans to enroll 23~116 subjects, and a phase 2 stage to explore efficacy, safety and tolerability of IBI3003 at RP2D in multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in Parts 1(dose escalation) & 2 (dose expansion) must satisfy all of the following criteria to be enrolled into the study:

  1. Age ≥18 years. For Part 1, age ≥18 years and ≤75 years.
  2. Documented initial diagnosis of multiple myeloma according to IMWG diagnostic criteria. Multiple myeloma is defined as clonal bone marrow plasma cells ≥10% or biopsy-proven bony or extramedullary plasmacytoma and any one or more of the following myeloma-defining events in protocol
  3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
  4. Life expectancy ≥3 months.
  5. Subjects with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol.

Exclusion Criteria:

1. Known active CNS involvement or exhibits clinical signs of meningeal involvement of multiple myeloma.
2. Have amyloidosis, plasma cell leukemia, Waldenstrom macroglobulinemia, POEMS syndrome, or solitary plasmacytoma, or smoldering MM as defined by the International Myeloma Working Group(IMWG) criteria.
3. Spinal cord compression that results in limited self-care occurs within 6 months prior to informed consent, or is expected to occur in the near future.
4. History of primary immunodeficiency.
5. Current or previous other malignancy within 3 years of study entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to 30 days post last dose
  Number of patients who Experienced related AEs from the first dose until 30 days after the last dose

SECONDARY OUTCOMES:
Dose limiting toxicities (DLTs) | Up to 28 days post first dose
  To evaluate the safety and tolerability of IBI3003

CONTACTS AND LOCATIONS:
Locations (13):
- Australia (3):
  - Wollongong Private Hospital, Wollongong, New South Wales
  - Austin Hospital, Heidelberg, Victoria
  - St Vincent's Hospital, Melbourne, Victoria
- China (10):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The first Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Tongji Medical College of HUST Tongji Hospital, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - ZhongShan Hospital FuDan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of XI'AN Jiaotong University, Xian, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No